CLINICAL TRIAL: NCT04954430
Title: The Reliability Assessment of Emergency Paramedics' Fatigue Using Automated Pupillometry
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-893
Record Dates: First submitted 2021-05-31; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-05

CONDITIONS: Mental Fatigue; Emergency Paramedics' Fatigue
Keywords: pupillary light reflex (PLR); automated quantitative pupillometry; Karolinska Sleepiness Scale (KSS); heart rate variability (HRV); electroencephalography (EEG)
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fatigue: After enrollments, subjects were assigned to perform mental fatigue-inducing experiment-a 90 min of monotonous simulated driving task. They underwent repeated measurements of quantitative pupillary light reflex (PLR) using an automated quantitative pupillometer at baseline and at an interval of 30 min during the task. Subjective ratings, heart rate variability (HRV), and electroencephalography (EEG) were performed simultaneously.
  Interventions: Diagnostic Test: pupillometer

INTERVENTIONS:
Diagnostic Test: pupillometer — The dynamic changes of PLR were measured using the PLR-3000 pupillometer (NeurOptics, CA, USA), a hand-held portable device. Determination of PLR with automated pupillometry can be performed with a rubber cup covering the measured eye and the subject's hand covering the non-measured eye. A flash of visible white light with a duration of 0.8 sec and a pulse intensity of 50 µW is delivered to induce a pupillary reflex, and repeated video images at more than 30 frames/sec are stored for 6.65 sec. The device provided the examiner with maximum and minimum pupil size (Init and End), constriction percentage (%PLR), latency (LAT), constriction and dilation velocity (CV and DV), and T75.

SUMMARY:
Due to the limitations of current approaches to assess emergency paramedics' fatigue, a portable, quick, easy, and objective technique is required to be developed. The aim of the study was to investigate the reliability of automated pupillometry to assess mental fatigue based on a driver simulator.

ELIGIBILITY:
Inclusion Criteria:

* All participants held valid driving license of more than 2 years, with at least half of a year driving experience, had regular sleep pattern, normal or corrected to normal vision and no history of any psychiatric disorder.

Exclusion Criteria:

* None.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy postgraduate students from Zhejiang University School of Medicine in China voluntarily participated in our study. All participants were asked to follow the below requirements before the tests: 1) refrain from alcohol, caffeine and tea within 12 h, 2) adequate sleep (almost 6~8 h) the day before, and 3) wash the hair within 24 h. Informed written consent and training were provided prior to entering the experiment.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
subjective assessments | Baseline
  Karolinska Sleepiness Scale (KSS), a 9-point scale for assessing sleepiness with responses ranging from extremely alert (1) to very sleepy (9) .
subjective assessments | 30 minutes
  Karolinska Sleepiness Scale (KSS), a 9-point scale for assessing sleepiness with responses ranging from extremely alert (1) to very sleepy (9) .
subjective assessments | 60 minutes
  Karolinska Sleepiness Scale (KSS), a 9-point scale for assessing sleepiness with responses ranging from extremely alert (1) to very sleepy (9) .
subjective assessments | 90 minutes
  Karolinska Sleepiness Scale (KSS), a 9-point scale for assessing sleepiness with responses ranging from extremely alert (1) to very sleepy (9) .
Standard deviation of the NN intervals of heart rate variability | Baseline
  Using the SA-3000P (Medicore, Korea) , subjects were instructed to stay with eyes open, be silent, and breath normally during measurement.
Standard deviation of the NN intervals of heart rate variability | 30 minutes
  Using the SA-3000P (Medicore, Korea) , subjects were instructed to stay with eyes open, be silent, and breath normally during measurement.
Standard deviation of the NN intervals of heart rate variability | 60 minutes
  Using the SA-3000P (Medicore, Korea) , subjects were instructed to stay with eyes open, be silent, and breath normally during measurement.
Standard deviation of the NN intervals of heart rate variability | 90 minutes
  Using the SA-3000P (Medicore, Korea) , subjects were instructed to stay with eyes open, be silent, and breath normally during measurement.
%PLR (percentage of change) | Baseline
  The dynamic changes of pupillary light reflex were measured using the PLR-3000 pupillometer (NeurOptics, CA, USA), a hand-held portable device. Determination of pupillary light reflex with automated pupillometry can be performed with a rubber cup covering the measured eye and the subject's hand covering the non-measured eye. A flash of visible white light with a duration of 0.8 sec and a pulse intensity of 50 µW is delivered to induce a pupillary reflex, and repeated video images at more than 30 frames/sec are stored for 6.65 sec.
%PLR (percentage of change) | 30 minutes
  The dynamic changes of pupillary light reflex were measured using the PLR-3000 pupillometer (NeurOptics, CA, USA), a hand-held portable device. Determination of pupillary light reflex with automated pupillometry can be performed with a rubber cup covering the measured eye and the subject's hand covering the non-measured eye. A flash of visible white light with a duration of 0.8 sec and a pulse intensity of 50 µW is delivered to induce a pupillary reflex, and repeated video images at more than 30 frames/sec are stored for 6.65 sec.
%PLR (percentage of change) | 60 minutes
  The dynamic changes of pupillary light reflex were measured using the PLR-3000 pupillometer (NeurOptics, CA, USA), a hand-held portable device. Determination of pupillary light reflex with automated pupillometry can be performed with a rubber cup covering the measured eye and the subject's hand covering the non-measured eye. A flash of visible white light with a duration of 0.8 sec and a pulse intensity of 50 µW is delivered to induce a pupillary reflex, and repeated video images at more than 30 frames/sec are stored for 6.65 sec.
%PLR (percentage of change) | 90 minutes
  The dynamic changes of pupillary light reflex were measured using the PLR-3000 pupillometer (NeurOptics, CA, USA), a hand-held portable device. Determination of pupillary light reflex with automated pupillometry can be performed with a rubber cup covering the measured eye and the subject's hand covering the non-measured eye. A flash of visible white light with a duration of 0.8 sec and a pulse intensity of 50 µW is delivered to induce a pupillary reflex, and repeated video images at more than 30 frames/sec are stored for 6.65 sec.

SECONDARY OUTCOMES:
Electroencephalography power in theta band | Baseline
  The eego™ mylab system (ANT Neuro, Germany) was applied to record the raw electroencephalography signal, using a 64-channel waveguard™ original electrode cap with electrodes in accordance with the international 10 ~ 20 Montage system. electroencephalography was sampled with a frequency of 1kHz using an eego™ amplifier. Electrode impedences of the selected channels were kept below 5 kΩ before recording.
Electroencephalography power in theta band | 30 minutes
  The eego™ mylab system (ANT Neuro, Germany) was applied to record the raw electroencephalography signal, using a 64-channel waveguard™ original electrode cap with electrodes in accordance with the international 10 ~ 20 Montage system. electroencephalography was sampled with a frequency of 1kHz using an eego™ amplifier. Electrode impedences of the selected channels were kept below 5 kΩ before recording.
Electroencephalography power in theta band | 60 minutes
  The eego™ mylab system (ANT Neuro, Germany) was applied to record the raw electroencephalography signal, using a 64-channel waveguard™ original electrode cap with electrodes in accordance with the international 10 ~ 20 Montage system. electroencephalography was sampled with a frequency of 1kHz using an eego™ amplifier. Electrode impedences of the selected channels were kept below 5 kΩ before recording.
Electroencephalography power in theta band | 90 minutes
  The eego™ mylab system (ANT Neuro, Germany) was applied to record the raw electroencephalography signal, using a 64-channel waveguard™ original electrode cap with electrodes in accordance with the international 10 ~ 20 Montage system. electroencephalography was sampled with a frequency of 1kHz using an eego™ amplifier. Electrode impedences of the selected channels were kept below 5 kΩ before recording.

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided